CLINICAL TRIAL: NCT04771546
Title: Evaluation of the Efficacy of an Intravaginal Treatment With Carboxymethyl-β-glucan and Polycarbophil on the Regression of Low-grade Cervical Intraepithelial Lesions
Brief Title: Efficacy of Intravaginal Carboxymethyl-β-glucan and Polycarbophil on Low-grade Cervical Lesions (GLUCANCIN)
Acronym: GLUCANCIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uriach Consumer Healthcare (Industry)
Collaborators: Hospital Universitario Infanta Leonor (Other); Hospital Universitario 12 de Octubre (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario Fundación Jiménez Díaz (Other); Hospital San Carlos, Madrid (Other); Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLUCANCIN V3 22/9/2020
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Human Papilloma Virus
Keywords: Human Papilomavirus; Cervical cancer; Low-grade Cervial intraepithelial lesions; High-Risk Papillomavirus; CIN1; beta-glucans
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Interventional, longitudinal, prospective, open label trial with a control group with randomized, consecutive recruitment for each group, to evaluate the safety and efficacy of carboxymethyl-beta-glucan and polycarbophil as a treatment for low-grade CIN associatedto HR-HPV infection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Colpofix) (Experimental): Intravaginal gel with Carboxymethyl-β-glucan and Polycarbophil
  Interventions: Device: Colpofix
- Control (No Intervention): No intervention (standard of care)

INTERVENTIONS:
Device: Colpofix — Intravaginal gel with carboxymtheyl beta-glucan and polycabophil. Posology: 1 application / day x 20 days, rest 10. Repeat 20 x 3 cycles
  Arms: Intervention (Colpofix)

SUMMARY:
A therapeutic strategy to neutralize the evasion mechanisms of HPV. Among these treatments are beta-glucans, polysaccharides of beta-D-glucose that, can influence the clearance of HPV. The objective of this study is to evaluate the efficacy of a gel with Carboxymethyl - β -Glucan and polycarbophil when applied intravaginally, on the regression of low-grade cervical intraepithelial lesions (CIN) associated to HR-HPV infection.

DETAILED DESCRIPTION:
Background

Human papillomavirus (HPV) infection represents a significant source of morbidity and mortality worldwide. High-risk oncogenic HPVs cause 99.7% of cervical cancers. 80% of sexually active women will be infected with HPV at some point in their life. Most of these infections are transitory and only if they are persistent and caused by a high-risk oncogenic HPV are they an important risk factor for the development of cervical intraepithelial lesions and invasive cervical cancer. Immunity plays a key factor in eliminating HPV infection. The innate immune response constitutes the first line of defense against infection during the early stages of infection, promoting a cytokine-mediated inflammatory response which links innate immunity with the adaptive immune response. HPV evasion of these immune defense mechanisms is critical for the persistence of the infection and leads to the development of preneoplastic lesions and ultimately to cervical cancer. One of most promising treatments is beta-glucans that seem capable of affecting the course of HPV infection, and consequently, the progression of its associated intraepithelial lesions.

Justification

β-glucans are a very diverse heterogeneous group of polysaccharides made up of D-glucose monomers linked by β-type glycosidic bonds.

β-glucans have been previously described in bacteria, fungi, yeasts (including brewer's yeast), plants and algae, where they play an important structural role in the cell wall or reservoir.

There are more than 6000 β-glucans studies. At least 4 receptors have been identified in mammals for the recognition of these molecules: lactosylceramide, scavengers, complement receptor 3 and dectin-1.

Commercial production of 1,3-β-glucans has been carried out by cultivating bacteria, yeasts, fungi, and plants.

Recent studies focusing on their influence on cytotoxic and helper T cells, APCs, inflammatory pathways, and oxidative burst (using reactive oxygen species to kill cells) have revealed that they may also have some anti-cancer properties. Some efforts have been made in the field of cervical cancer prevention and it has been shown that β-glucans can also affect HPV infection. Carboxymethyl β-glucan gel treatment was studied in a group of affected individuals by CIN1. This case-control study demonstrated that it has an anti-cervical cancer role in CIN1 regression. In 2010, two studies were conducted on the topic of "the influence of β-glucans" on HPV-related lesions in the genital area. "The first study found that β-glucans can treat infection-related lesions and the second study revealed the efficacy of beta-glucan treatment for HPVCIN1 lesions. These studies suggested that, in addition to the anticancer effects of beta-glucans, they also have some effects on infection by HPV, the main cause of cervical cancer.

On the other hand, the local treatment of vaginal problems has been known since ancient times, and more recently it has been favored over oral treatments due to the achievement of higher local concentrations of drugs and fewer interactions of the active principles and interference with the gastrointestinal tract. Vaginal products are marketed in the form of tablets, capsules, pessaries or ovules and semisolid forms (creams, ointments and gels), being available as products for the treatment and prevention of vaginal infections. Conventional dosage forms are associated with poor distribution and retention, primarily due to the self-cleaning action of the vagina. Among the commercialized dosage forms, semisolids, in particular gels, have been considered the preferred ones as they spread easily over the vaginal surface area. Additionally, due to their high water content, they confer moisture and lubrication effects that help alleviate the symptoms of conditions associated with vaginal dryness.

Bioadhesion refers to the binding of natural or synthetic macromolecules to a biological tissue. Mucoadhesion is considered a particular case of bioadhesion whenever the binding occurs with mucous glycoproteins (mucin) or mucous membranes. The translation of these concepts into pharmaceutical technology has been widely studied through the use of bioadhesive polymers. Among the most used in vaginal formulations are polyacrylates (such as carbomers and polycarbophils), cellulose derivatives (hydroxyethylcellulose (HEC), hydroxypropylcellulose (HPC), hydroxypropylmethylcellulose (HPMC), etc.), chitosan, hyaluronic acid and its derivatives, starch, pectin, natural gums and sodium alginate. In addition to increasing the retention time of vaginal formulations, thus promoting therapeutic duration and efficacy and improving patient comfort and adherence, these excipients also allow controlled drug release, thus improving local pharmacokinetics.

Polycarbophil and carbomer (polyacrylate) vaginal applications have been specially studied in vitro and in vivo, and have been included in various proprietary formulations as well as actual marketed products. These polymers have the additional advantage of being acidic, allowing the correction and maintenance of vaginal pH, and their acid-buffering capacity has been explored as a strategy for the treatment of bacterial vaginosis and the prevention of vaginosis recurrence for prevent the proliferation of pathogens, while promoting the restoration of the protective flora of Lactobacillus.

Polycarbophil, in particular, has been widely used for its bioadhesive properties, especially after a 1-3% polycarbophil gel was shown to maintain vaginal acidity for 3-4 days after a single application in postmenopausal women and A polycarbophil-carbomer vaginal gel was proven in women with suspected and confirmed bacterial vaginosis to show a reduction in vaginal pH in both trials, and a high clinical cure rate in confirmed vaginosis cases compared to placebo.

The objective of this study is to evaluate the efficacy of a gel with Carboxymethyl - β -Glucan and polycarbophil when applied intravaginally on the regression of low-grade Cervical intraepithelial lesions (CIN) associated to HR-HPV infection.

ELIGIBILITY:
Inclusion Criteria:

* Woman between 30 and 50 years old
* Capable of understanding the Pacient Information Sheet and the Informed Consent form
* Accepting her particpation in the study and signing the Informed Consent
* LSIL/CIN1 hystological result on cervical biopsy preceeded by HR-HPV+ test (genotypes 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68)
* Cervical cytology ≥ ASCUS or precceded by a HPV16+ test and negative cervical cytology for lesion or malignancy but with CIN1 colposcopy and biopsy.

Exclusion Criteria:

* Cervical cytology suspicious of invasive cervical cancer
* Current or previous pregnancy ended before six weeks in relation to the start of the study.
* Vaccination against HPV.
* Clinically relevant pathology linked to immunodeficiency.
* Immunosuppressive treatment active or finished before six months in relation to the start of the study. In the specific case of corticosteroids, all women who are receiving corticosteroid treatment currently or recently (defined as the two weeks prior to the start of the study) or if she has received 2 or more cycles of corticosteroids in equal or greater than 20 mg / day of predsinone (or equivalent) orally or parenterally, for one week duration at least in the year prior to the start of the study. The use of inhaled corticosteroids, Nasal or topical are not exclusion criteria.
* Undiagnosed abnormal genital bleeding.
* Total hysterectomy.
* Presence of genital warts and other symptomatic vulvovaginal infections.
* Documented history of cervical pathology caused by HPV.
* Current systemic and / or gynecological disease that contraindicates the use of Colpofix.
* Contraindications to the use of Colpofix or known allergies to any of its components
* Simultaneous participating in a clinical study of an investigational drug or that could interfere with the use of Colpofix.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in CIN1 regression rate | 24 months (6, 12, 18 and 24 months)
  CIN evaluation by biopsy

SECONDARY OUTCOMES:
CIN1 lesion regression or clearance time | 24 months (6, 12, 18 and 24 months)
  CIN evaluation by biopsy
Progression to CIN2+ rate | 24 months (6, 12, 18 and 24 months)
  CIN evaluation by biopsy
HPV clearance rate | 24 months (6, 12, 18 and 24 months)
  Evaluation of HPV clearance time by HPV PCR test
HPV clearance time | 24 months (6, 12, 18 and 24 months)
  Evaluation of HPV clearance time by HPV PCR test
Normalization rate of abnormal cytology | 24 months (6, 12, 18 and 24 months)
  Evaluation of normal/abnormal cytologies
Normalization time of abnormal cytology | 24 months (6, 12, 18 and 24 months)
  Evaluation of normal/abnormal cytologies
Normalization rate of abnormal colposcopy | 24 months (6, 12, 18 and 24 months)
  Evaluation of normal/abnormal colposcopy
Normalization time of abnormal colposcopy | 24 months (6, 12, 18 and 24 months)
  Evaluation of normal/abnormal colposcopy

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Hernández Aguado, MD, Principal Investigator — Hospital Universitario Infanta Leonor
Locations (5):
- Spain (5):
  - Hospital Universitario Infanta Leonor, Vallecas, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geller A, Shrestha R, Yan J. Yeast-Derived beta-Glucan in Cancer: Novel Uses of a Traditional Therapeutic. Int J Mol Sci. 2019 Jul 24;20(15):3618. doi: 10.3390/ijms20153618. PMID 31344853
- [Background] Chaichian S, Moazzami B, Sadoughi F, Haddad Kashani H, Zaroudi M, Asemi Z. Functional activities of beta-glucans in the prevention or treatment of cervical cancer. J Ovarian Res. 2020 Mar 5;13(1):24. doi: 10.1186/s13048-020-00626-7. PMID 32138756
- [Background] Stentella P, Biamonti A, Carraro C, Inghirami P, Mancino P, Pietrangeli D, Votano S, Lazzari P, DE Medici C. Efficacy of carboxymethyl beta-glucan in cervical intraepithelial neoplasia: a retrospective, case-control study. Minerva Ginecol. 2017 Oct;69(5):425-430. doi: 10.23736/S0026-4784.17.04053-9. PMID 28675291
- [Background] Pietrantoni E, Signore F, Berardi G, Donadio F, Donadio C. [Role of beta-glucan in the treatment of recurrent candidiasis and HPV-correlated lesions and reparative process of epidermis]. Minerva Ginecol. 2010 Feb;62(1):1-5. Italian. PMID 20186110
- [Background] Scardamaglia P, Carraro C, Mancino P, Stentella P. [Effectiveness of the treatment with beta-glucan in the HPV-CIN 1 lesions]. Minerva Ginecol. 2010 Oct;62(5):389-93. Italian. PMID 20938424
- [Background] Palmeira-de-Oliveira R, Palmeira-de-Oliveira A, Martinez-de-Oliveira J. New strategies for local treatment of vaginal infections. Adv Drug Deliv Rev. 2015 Sep 15;92:105-22. doi: 10.1016/j.addr.2015.06.008. Epub 2015 Jul 2. PMID 26144995
- [Background] Fiorilli A, Molteni B, Milani M. Successful treatment of bacterial vaginosis with a policarbophil-carbopol acidic vaginal gel: results from a randomised double-blind, placebo-controlled trial. Eur J Obstet Gynecol Reprod Biol. 2005 Jun 1;120(2):202-5. doi: 10.1016/j.ejogrb.2004.10.011. PMID 15925053